CLINICAL TRIAL: NCT05235867
Title: Secretin Levels in Refeeding-induced Polyuria (Cross Section)
Brief Title: Secretin in Refeeding
Status: Recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Elaine L. Rosen, MD, Principal Investigator, University of California, Los Angeles
Other Study IDs: IRB#21-001489
Record Dates: First submitted 2022-02-01; First posted 2022-02-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Anorexia in Adolescence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dumpers: * male and female patients
  * age 13-24 years
  * diagnosis of restrictive-type anorexia nervosa
  * hospitalization for nutritional support
  * >4 cc/kg/day of urine output (a.k.a. "fluid dumpers"; n=5)
- non-dumpers: * male and female patients
  * age 13-24 years
  * diagnosis of restrictive-type anorexia nervosa
  * hospitalization for nutritional support
  * <2 cc/kg/d of urine output (a.k.a. "non-dumpers"; n=5)

SUMMARY:
Patients with restrictive-type anorexia nervosa who are admitted to the hospital for feeding often urinate excessive amounts. Others have changes in the way that they handle acid and base. These issues prolong hospitalizations. Current data suggest that one hormone--named secretin--may control both urine output and how the body handles acid and base. This study will evaluate whether secretin levels are different in anorexic patients who urinate an excessive amount compared to those who urinate normal amounts. For this study, patients will have one extra blood draw before and after one meal during their hospitalization. The blood draw before the meal coincides with a standard of care blood draw. Also after the meal, subjects will be asked to provide one extra urine sample. Information from subject's medical records will also be used.

ELIGIBILITY:
Inclusion Criteria:

* Group 1:

  * male and female patients
  * age 13-24 years
  * diagnosis of restrictive-type anorexia nervosa
  * hospitalization for nutritional support
  * >4 cc/kg/day of urine output (a.k.a. "fluid dumpers"; n=5)
* Group 2:

  * male and female patients
  * age 13-24 years
  * diagnosis of restrictive-type anorexia nervosa
  * hospitalization for nutritional support
  * <2 cc/kg/d of urine output (a.k.a. "non-dumpers"; n=5)

Exclusion Criteria:

* 5150 hold
* Anti-depressant, anti-psychotic, or anticonvulsant medications
* Previous hospitalization within the past 6 months
* Underlying metabolic disorder not related to anorexia nervosa (including chronic kidney disease, renal tubular disorders, and underlying endocrine disorders)
* Pregnancy
* NG or G-tube feeds after day 2 of hospitalization
* > 10% of nutritional needs from supplemental feeds

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents with restrictive-type anorexia hospitalized for medical nutritional stabilization.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in secretin | 1 hour
  Change in secretin value from pre- to post- meal

SECONDARY OUTCOMES:
Change in serum bicarbonate | 1 hour
  Change in bicarbonate value from pre- to post- meal

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles (UCLA), Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No